CLINICAL TRIAL: NCT07016880
Title: The Effect of Virtual Reality Intervention on Preoperative Anxiety, Physiological Parameters and Patient Satisfaction in Women Scheduled for Gynecological Oncology Surgery: A Randomised Controlled Trial
Brief Title: Anxiety, Physiological Parameters, Patient Satisfaction and VR in Gynecological Oncology Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Uslu Sahan, Associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/93
Record Dates: First submitted 2025-05-21; First posted 2025-06-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Preoperative Anxiety; Women's Health; Gynecological Cancers; Gynecological Surgery
Keywords: Gynecological Surgery; Gynecological Oncology; Preoperative Anxiety; Preoperative Anxiety Management; Virtual Reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Participants in this group will receive a virtual reality intervention before surgery. Anxiety, physiological parameters, and satisfaction will be assessed both before and after the VR session.
  Interventions: Behavioral: Virtual Reality Relaxation Session
- Standard Care Group (No Intervention): Participants in this group will receive standard preoperative care. The same measurements will be taken before and after standard care.

INTERVENTIONS:
Behavioral: Virtual Reality Relaxation Session — A 20 minute virtual reality session using visual and auditory stimuli for relaxation before surgery. Delivered via VR headset.
  Arms: Virtual Reality Group

SUMMARY:
Surgical procedures often cause significant anxiety in patients, particularly among women undergoing gynecological oncology surgeries. Preoperative anxiety is a common and preventable condition that can negatively affect both physiological parameters and the overall surgical experience. It may lead to increased heart rate, elevated blood pressure, respiratory distress, and psychological discomfort, increasing the risk of complications during and after surgery. Women facing gynecological cancer surgery often experience heightened anxiety due to concerns about survival, loss of reproductive organs, body image changes, and sexual health.

Virtual reality (VR) has emerged as a promising non-pharmacological approach for reducing preoperative anxiety. By immersing patients in a calming virtual environment that engages visual and auditory senses, VR helps promote relaxation, reduce stress, and enhance the patient's sense of control before surgery. It is safe, easy to implement, cost-effective, and does not have the side effects associated with medications.

Although VR has demonstrated effectiveness in reducing anxiety in various surgical contexts-including orthopedic, colorectal, and minor gynecological procedures-its impact in gynecologic oncology surgery remains underexplored. This randomized controlled trial aims to evaluate the effect of a VR intervention on preoperative anxiety, physiological parameters (blood pressure, heart rate, respiratory rate, oxygen saturation), and patient satisfaction in women scheduled for gynecologic oncology surgery.

Participants will be randomly assigned to either the intervention group (receiving VR) or the control group (receiving standard care). Anxiety and physiological measures will be evaluated before and after the respective intervention in both groups. Patient satisfaction will be assessed once, immediately after the intervention and before surgery.

The primary objective is to assess whether VR effectively reduces preoperative anxiety and stabilizes physiological indicators. The secondary objective is to evaluate patient satisfaction with the preoperative experience. This study will contribute to the evidence base for using VR as a nursing-led, non-invasive strategy to enhance surgical care in gynecologic oncology.

DETAILED DESCRIPTION:
Preoperative anxiety is a common and preventable psychological condition that significantly affects surgical outcomes and patient well-being. Women undergoing gynecologic oncology surgery often face elevated levels of anxiety due to the severity of their diagnosis, potential loss of reproductive organs, and concerns related to survival, body image, and sexuality. These psychological stressors can lead to physiological changes such as increased blood pressure, heart rate, and respiratory distress, which in turn may complicate surgical procedures and recovery. Managing preoperative anxiety effectively is essential not only to minimize surgical risk but also to improve patient satisfaction and postoperative adaptation.

Pharmacological methods used to manage preoperative anxiety can carry risks such as side effects, drug interactions, and delayed postoperative recovery. For this reason, non-pharmacological interventions such as virtual reality (VR) have gained popularity in recent years. VR allows patients to be immersed in a multisensory virtual environment that helps distract their attention away from surgery-related fears and fosters relaxation. Studies in orthopedic, colorectal, and minor gynecologic procedures have shown that VR can reduce anxiety and improve physiological responses before surgery. However, limited evidence exists regarding its use in women undergoing gynecologic oncology surgery-a population that faces unique psychological and physical challenges.

This study is a two-arm randomized controlled trial designed to evaluate the effectiveness of a virtual reality (VR) intervention in reducing preoperative anxiety and stabilizing physiological parameters in women scheduled for gynecologic oncology surgery via laparotomy. A total of 66 participants will be randomly assigned to either the intervention group (VR session) or the control group (standard care). In both groups, anxiety levels and physiological parameters (blood pressure, heart rate, respiratory rate, and oxygen saturation) will be assessed before and after the intervention. Patient satisfaction with preoperative care will be assessed only once, following the intervention or standard care session, immediately before surgery.

Eligibility criteria include adult women (≥18 years) with a confirmed diagnosis of gynecologic cancer who are aware of their diagnosis and scheduled for their first surgical intervention via laparotomy. Participants must have an ECOG Performance Status ≤2 and must not have any cognitive, visual, auditory, or psychiatric impairments that could interfere with communication or VR use. Exclusion criteria include recurrent cancer, motion sensitivity (e.g., vertigo or migraines), or any condition preventing the use of VR headsets.

The study aims to contribute new evidence supporting the use of VR as a nurse-led, low-risk, and effective non-pharmacological approach to improve preoperative experiences and perioperative outcomes in women facing gynecologic oncology surgery.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have a confirmed diagnosis of gynecological cancer.
* The participant must be aware of their gynecological cancer diagnosis.
* Participants must be 18 years of age or older.
* Verbal and written informed consent to participate in the study must be obtained.
* The participant must be able to communicate verbally and in writing in Turkish.
* No communication impairments (e.g., visual, auditory, or cognitive) should be present.
* This must be the participant's first surgical intervention related to gynecological oncology.
* Eastern Cooperative Oncology Group (ECOG) Performance Status must not exceed 2.
* The planned surgical procedure must be a laparotomy.

Exclusion Criteria:

* History of recurrent gynecological cancer.
* Presence of vision problems that prevent the use of VR goggles, including participants who wear glasses or have uncorrected vision impairment.
* Presence of conditions such as migraines, vertigo, active nausea, vomiting, or frequent headaches.
* Sensitivity to motion sickness.
* Diagnosis of a psychiatric condition, whether under pharmacological or non-pharmacological treatment.
* Withdrawal of consent during the study.
* Removal of the virtual reality headset during the intervention.
* Development of any medical complications during the intervention period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Score | Immediately before and immediately after the intervention, on the day of surgery
  Change in anxiety levels as measured by the State-Trait Anxiety Inventory - State subscale (STAI-S), a 20-item scale ranging from 20 to 80. Higher scores indicate greater anxiety.
Change in Systolic and Diastolic Blood Pressure | Immediately before and immediately after the intervention, on the day of surgery
  Change in systolic and diastolic blood pressure measured in mmHg, recorded using a calibrated automated monitor.
Change in Heart Rate | Immediately before and immediately after the intervention, on the day of surgery
  Change in heart rate measured in beats per minute (bpm), recorded using standard physiological monitoring equipment.
Change in Respiratory Rate | Immediately before and immediately after the intervention, on the day of surgery
  Change in respiratory rate recorded in breaths per minute using standard clinical observation.
Change in Peripheral Oxygen Saturation | Immediately before and immediately after the intervention, on the day of surgery
  Change in oxygen saturation levels (%) measured using pulse oximetry.

SECONDARY OUTCOMES:
Preoperative Patient Satisfaction Score | Immediately after the intervention (same day, pre-surgery)
  Patient satisfaction will be assessed using a Visual Analog Scale (VAS), ranging from 0 to 10, where zero indicates 'Not satisfied at all' and 10 indicates 'Extremely satisfied.' Participants will be asked to rate their overall satisfaction with the care they received throughout the preoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Uslu Sahan, Assoc Prof, Principal Investigator — Hacettepe University Faculty of Nursing
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koo CH, Park JW, Ryu JH, Han SH. The Effect of Virtual Reality on Preoperative Anxiety: A Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Sep 29;9(10):3151. doi: 10.3390/jcm9103151. PMID 33003411
- [Result] Vogt L, Klasen M, Rossaint R, Goeretz U, Ebus P, Sopka S. Virtual Reality Tour to Reduce Perioperative Anxiety in an Operating Setting Before Anesthesia: Randomized Clinical Trial. J Med Internet Res. 2021 Sep 1;23(9):e28018. doi: 10.2196/28018. PMID 34252034
- [Result] Asiri S, Guilhermino M, Duff J. The effectiveness of using virtual reality technology for perioperative anxiety among adults undergoing elective surgery: a randomised controlled trial protocol. Trials. 2022 Dec 2;23(1):972. doi: 10.1186/s13063-022-06908-3. PMID 36461040
- [Result] Turrado V, Guzman Y, Jimenez-Lillo J, Villegas E, de Lacy FB, Blanch J, Balibrea JM, Lacy A. Exposure to virtual reality as a tool to reduce peri-operative anxiety in patients undergoing colorectal cancer surgery: a single-center prospective randomized clinical trial. Surg Endosc. 2021 Jul;35(7):4042-4047. doi: 10.1007/s00464-021-08407-z. Epub 2021 Mar 8. PMID 33683433